CLINICAL TRIAL: NCT00746330
Title: A Randomized, Double-blind, Double-dummy, Multi-centre, 4-way Cross-over Study to Compare the Single Dose Bronchodilatory Effect of Formoterol Fumarate in Combination With Mometasone Furoate Delivered Via Pressurized Metered Dose Inhaler (pMDI) to Placebo Delivered Via pMDI in Children Aged 5-11 Years Old With Persistent Asthma
Brief Title: Single Dose Study of the Effect of Formoterol Fumarate in Combination With Mometasone Furoate Inhaled Via a Pressurized Metered Dose Inhaler (pMDI) in Children Aged 5-11 Years Old With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMFF258C2204
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Asthma; Children; Persistent asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- F12M - PL - F12D - MFF (Experimental): Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 2: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 3: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 4: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
  Interventions: Drug: Mometasone furoate/formoterol fumarate (MFF); Drug: Formoterol fumarate 12 μg pMDI (F12M); Drug: Formoterol fumarate 12 μg DPI (F12D); Drug: Placebo to F12D; Drug: Placebo to F12M/MFF
- F12D - F12M - MFF - PL (Experimental): Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 2: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 3: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 4: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
  Interventions: Drug: Mometasone furoate/formoterol fumarate (MFF); Drug: Formoterol fumarate 12 μg pMDI (F12M); Drug: Formoterol fumarate 12 μg DPI (F12D); Drug: Placebo to F12D; Drug: Placebo to F12M/MFF
- MFF - F12D - PL - F12M (Experimental): Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 2: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 3: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 4: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
  Interventions: Drug: Mometasone furoate/formoterol fumarate (MFF); Drug: Formoterol fumarate 12 μg pMDI (F12M); Drug: Formoterol fumarate 12 μg DPI (F12D); Drug: Placebo to F12D; Drug: Placebo to F12M/MFF
- PL - MFF - F12M - F12D (Experimental): Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 2: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 3: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 4: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
  Interventions: Drug: Mometasone furoate/formoterol fumarate (MFF); Drug: Formoterol fumarate 12 μg pMDI (F12M); Drug: Formoterol fumarate 12 μg DPI (F12D); Drug: Placebo to F12D; Drug: Placebo to F12M/MFF

INTERVENTIONS:
Drug: Mometasone furoate/formoterol fumarate (MFF) — Formoterol fumarate dihydrate / mometasone furoate combination product 10 μg / 100 μg delivered via Pressurized Metered Dose Inhaler (pMDI). One dose consisted of 2 puffs x 5 μg / 50 μg.
Drug: Formoterol fumarate 12 μg pMDI (F12M) — Formoterol fumarate dihydrate 12 μg delivered via Pressurized Metered Dose Inhaler (pMDI) (1 dose = 2 puffs x 6 μg).
Drug: Formoterol fumarate 12 μg DPI (F12D) — Formoterol fumarate dihydrate 12 μg delivered via Dry Powder Inhaler (DPI).
Drug: Placebo to F12D — Placebo to formoterol fumarate DPI delivered via DPI
Drug: Placebo to F12M/MFF — Placebo to formoterol fumarate pMDI and formoterol fumarate / mometasone furoate delivered via pMDI

SUMMARY:
This study is being conducted to compare the pharmacodynamics (bronchodilation, onset and duration of action), of a single dose of formoterol fumarate in combination with mometasone furoate to placebo in children of 5-11 years with persistent asthma. The study will also assess the bronchodilatory effect of a single dose of formoterol fumarate alone and in combination with mometasone furoate delivered via a pressurized metered dose inhaler (pMDI) to the bronchodilatory effect of formoterol fumarate delivered via a dry powder inhaler (DPI). Furthermore, pharmacokinetic assessments of plasma and urine will also be conducted throughout the study to assess systemic exposure following administration of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 11 years of age of either sex and of any race
* A diagnosis (according to the Global Initiative for Asthma [GINA] guidelines) of persistent asthma for a period of at least 6 months prior to screening and must have been on a stable asthma regimen (daily dose unchanged) for at least 4 weeks prior to screening
* β2-agonist reversibility, defined as an increase in absolute FEV1 of ≥12% within 30 minutes after administration of 200μg of salbutamol without the use of a spacer or its equivalent in accordance with ATS/ERS standards
* A child must have an FEV1 of ≥ 60% and ≤ 90% of Polgar predicted when all restricted medications have been withheld for the appropriate intervals

Exclusion Criteria:

* Use of other investigational drugs at the time of enrolment, or within 30 days or 5 half-lives of enrolment, whichever is longer.
* History of malignancy of any organ system within past 5 years.
* Pre-dose change (increase or decrease) in absolute FEV1 of 15% at Visit 2, compared with value at screening.
* Hospitalized or had an emergency room treatment for an acute asthma exacerbation in the 1 month prior to Visit 1, or who had a clinical deterioration of asthma between Visits 1 and 2 that resulted in emergency treatment, hospitalization, or treatment with excluded asthma medication.
* Significant medication condition or situation.
* QTc > 440 msec (boys) or > 450 msec (girls) on electrocardiogram(ECG) assessment at screening.
* Upper or lower respiratory tract infection within 4 weeks prior to screening.
* Chronic conditions affecting the respiratory tract or chronic lung diseases.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Oklahoma City, Oklahoma
- Colombia (2):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Lima, Peru

RESULTS

PARTICIPANT FLOW:
Groups:
- F12M, PL, F12D, MFF: Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Formoterol fumarate 12 μg via Pressurized Metered Dose Inhaler (pMDI) + placebo to formoterol fumarate via Dry Powder Inhaler (DPI); Period 2: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 3: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 4: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
- F12D, F12M, MFF, PL: Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 2: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 3: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 4: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
- MFF, F12D, PL, F12M: Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 2: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 3: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 4: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
- PL, MFF, F12M, F12D: Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 2: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI; Period 3: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 4: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
Period: Period 1
Arm/Group | F12M, PL, F12D, MFF | F12D, F12M, MFF, PL | MFF, F12D, PL, F12M | PL, MFF, F12M, F12D
Started | 7 | 9 | 9 | 7
Completed | 7 | 9 | 8 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Abnormal test procedure result | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | F12M, PL, F12D, MFF | F12D, F12M, MFF, PL | MFF, F12D, PL, F12M | PL, MFF, F12M, F12D
Started | 7 | 9 | 8 | 7
Completed | 7 | 9 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | F12M, PL, F12D, MFF | F12D, F12M, MFF, PL | MFF, F12D, PL, F12M | PL, MFF, F12M, F12D
Started | 7 | 9 | 8 | 7
Completed | 7 | 9 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | F12M, PL, F12D, MFF | F12D, F12M, MFF, PL | MFF, F12D, PL, F12M | PL, MFF, F12M, F12D
Started | 7 | 9 | 8 | 7
Completed | 7 | 9 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- F12M, PL, F12D, MFF: Participants received a single dose of each treatment in the following order, separated by a washout period of 6-7 days: Period 1: Formoterol fumarate 12 μg via pMDI + placebo to formoterol fumarate via DPI; Period 2: Placebo to formoterol fumarate / mometasone furoate via pMDI + placebo to formoterol fumarate via DPI; Period 3: Placebo to formoterol fumarate / mometasone furoate via pMDI + formoterol fumarate via DPI; Period 4: Formoterol fumarate / mometasone furoate 10 μg / 100 μg via pMDI + placebo to formoterol fumarate via DPI. Participants were allowed to continue their regular asthma maintenance inhaled corticosteroid medication throughout the study and were supplied with the short-acting β2-agonist (SABA) salbutamol as rescue medication.
- Total: Total of all reporting groups
Arm/Group | F12M, PL, F12D, MFF | F12D, F12M, MFF, PL | MFF, F12D, PL, F12M | PL, MFF, F12M, F12D | Total
Number analyzed (Participants) | 7 | 9 | 9 | 7 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 9 | 9 | 7 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.63) | 9.4 (1.51) | 7.9 (1.83) | 10.1 (1.21) | 9.1 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 4 | 17
  Male | 5 | 3 | 4 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 2 | 11
  Not Hispanic or Latino | 5 | 7 | 4 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 3
  White | 5 | 4 | 3 | 4 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Standardized Forced Expiratory Volume in 1 Second (FEV1) Using Area Under the Curve (AUC) From 0 to 12 Hours (0-12h) Post-dose by Treatment
Description: For FEV1 AUC(0-12h) the trapezoidal rule was applied using planned time measurements to calculate the AUC up to and including the last measurement recorded before intake of rescue medication. The AUC was standardized by dividing by the length of time for which measurements of FEV1 were included in the calculation of the AUC thus adjusting for subjects who were unable to complete the measurements during the 12-hour observation period and without inhaling rescue medication. The unit of the AUC was in L, being a weighted average of the acceptable FEV1 measurements recorded over 12 hours post dose
Time Frame: From 0 to 12 Hours (0-12h) post-dose, after each treatment administered (approximately 1 treatment a week for 4 weeks of treatment).
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Groups:
- MFF10: Formoterol fumarate 10μg/Mometasone furoate 100μg via pMDI
- F12M: Formoterol fumarate 12 μg via pMDI/ Placebo via DPI
- F12D: Placebo via pMDI/ Formoterol fumarate 12 μg via DPI
- Placebo: Placebo via pMDI/ Placebo via DPI
Arm/Group | MFF10 | F12M | F12D | Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 31
liters | 1.77 (.042) [1.69 to 1.86] | 1.77 (.042) [1.69 to 1.85] | 1.80 (.042) [1.72 to 1.89] | 1.71 (.042) [1.62 to 1.79]

2. Secondary Outcome: Serial FEV1 Measurement (i.e. at 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose) Following Inhalation of a Single Dose of Study Medication to Evaluate the Onset and Duration of the Bronchodilatory Effect
Description: All efficacy evaluations were based on spirometry assessments of lung function. FEV1 is the maximum amount of air expired in one second. At Visits 2, 3, 4 and 5, spirometry assessments were performed in the clinic at predose and again at 5 and 30 minutes and 1, 2, 4, 8 and 12 hours post-dose within ± 5 minutes of the scheduled time for the time points up to and including 60 minutes post-dose and then within ± 10 minutes for all subsequent time points. Spirometry equipment and performance of spirometric testing were in accordance with the (ATS / ERS) standards.
Time Frame: 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | MFF10 | F12M | F12D | Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 31
liters
  5 minutes | 1.74 [1.70 to 1.79] | 1.77 [1.72 to 1.81] | 1.77 [1.73 to 1.82] | 1.68 [1.63 to 1.72]
  30 minutes | 1.79 [1.75 to 1.84] | 1.80 [1.75 to 1.85] | 1.82 [1.77 to 1.87] | 1.69 [1.64 to 1.74]
  1 hour (N=32, 31, 29, 31) | 1.81 [1.75 to 1.87] | 1.80 [1.74 to 1.86] | 1.86 [1.79 to 1.92] | 1.72 [1.66 to 1.78]
  2 hours | 1.81 [1.74 to 1.87] | 1.79 [1.72 to 1.85] | 1.85 [1.79 to 1.91] | 1.73 [1.67 to 1.79]
  4 hours | 1.81 [1.73 to 1.88] | 1.79 [1.71 to 1.87] | 1.84 [1.76 to 1.92] | 1.72 [1.64 to 1.80]
  8 hours | 1.76 [1.69 to 1.83] | 1.75 [1.69 to 1.82] | 1.79 [1.72 to 1.86] | 1.70 [1.63 to 1.77]
  12 hours | 1.72 [1.67 to 1.78] | 1.71 [1.65 to 1.76] | 1.76 [1.70 to 1.81] | 1.66 [1.61 to 1.72]

3. Secondary Outcome: Serial Forced Vital Capacity (FVC) Measurement (i.e. at 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose) Following Inhalation of a Single Dose of Study Medication to Evaluate the Onset and Duration of the Bronchodilatory Effect
Description: All efficacy evaluations were based on spirometry assessments of lung function. FVC is the volume (liters) of air that can forcibly be blown out after full inspiration. At Visits 2, 3, 4 and 5, spirometry assessments were performed in the clinic at predose and again at 5 and 30 minutes and 1, 2, 4, 8 and 12 hours post-dose within ± 5 minutes of the scheduled time for the time points up to and including 60 minutes post-dose and then within ± 10 minutes for all subsequent time points. Spirometry equipment and performance of spirometric testing were in accordance with the ATS / ERS standards.
Time Frame: 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | MFF10 | F12M | F12D | Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 31
liters
  5 minutes | 2.09 [2.04 to 2.14] | 2.09 [2.05 to 2.14] | 2.09 [2.04 to 2.13] | 2.08 [2.03 to 2.13]
  30 minutes | 2.12 [2.07 to 2.17] | 2.11 [2.06 to 2.16] | 2.11 [2.06 to 2.16] | 2.08 [2.03 to 2.13]
  1 hour (N=32, 31, 29, 31) | 2.14 [2.09 to 2.20] | 2.09 [2.03 to 2.14] | 2.15 [2.09 to 2.21] | 2.10 [2.04 to 2.15]
  2 hours | 2.11 [2.05 to 2.17] | 2.08 [2.02 to 2.14] | 2.14 [2.08 to 2.20] | 2.11 [2.05 to 2.17]
  4 hours | 2.12 [2.06 to 2.17] | 2.08 [2.02 to 2.14] | 2.12 [2.07 to 2.18] | 2.11 [2.05 to 2.17]
  8 hours | 2.09 [2.04 to 2.15] | 2.09 [2.04 to 2.15] | 2.10 [2.04 to 2.15] | 2.09 [2.04 to 2.15]
  12 hours | 2.07 [2.01 to 2.13] | 2.05 [1.99 to 2.11] | 2.09 [2.03 to 2.15] | 2.06 [2.00 to 2.12]

4. Secondary Outcome: Serial Peak Expiratory Flow Rate (PEF) Measurement (i.e. at 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose) Following Inhalation of a Single Dose of Study Medication to Evaluate the Onset and Duration of the Bronchodilatory Effect
Description: All efficacy evaluations were based on spirometry assessments of lung function. PEF is the greatest airflow rate achieved during forced exhalation with lungs fully inflated. At Visits 2, 3, 4 and 5, spirometry assessments were performed in the clinic at predose and again at 5 and 30 minutes and 1, 2, 4, 8 and 12 hours post-dose within ± 5 minutes of the scheduled time for the time points up to and including 60 minutes post-dose and then within ± 10 minutes for all subsequent time points. Spirometry equipment and performance of spirometric testing were in accordance with the ATS/ERS standards
Time Frame: 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | MFF10 | F12M | F12D | Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 31
liters
  5 minutes | 246.65 [238.31 to 254.99] | 248.17 [239.72 to 256.63] | 250.05 [241.48 to 258.62] | 237.85 [229.40 to 246.30]
  30 minutes | 255.69 [245.56 to 265.81] | 253.37 [243.14 to 263.59] | 257.81 [247.48 to 268.14] | 243.59 [233.36 to 253.82]
  1 hour (N=32, 31, 29, 31) | 261.18 [250.97 to 271.38] | 257.08 [246.79 to 267.38] | 262.95 [252.47 to 273.43] | 248.24 [237.94 to 258.54]
  2 hours | 261.45 [250.74 to 272.17] | 259.28 [248.45 to 270.10] | 267.91 [256.98 to 278.84] | 248.88 [238.05 to 259.70]
  4 hours | 264.68 [253.09 to 276.26] | 258.92 [247.24 to 270.60] | 265.20 [253.42 to 276.98] | 249.07 [237.39 to 260.76]
  8 hours | 257.96 [246.21 to 269.72] | 255.27 [247.41 to 267.12] | 262.61 [250.65 to 274.56] | 248.47 [236.61 to 260.33]
  12 hours | 255.48 [243.94 to 267.02] | 250.71 [239.06 to 262.37] | 259.71 [248.05 to 271.37] | 244.13 [232.59 to 255.66]

5. Secondary Outcome: Plasma Formoterol Concentrations (Pmol/L) Following a Single Dose of Formoterol Fumarate Alone and in Combination With Mometasone Furoate Via the pMDI and Formoterol Fumarate Via the Dry Powder Inhaler (DPI)
Description: Unchanged racemic formoterol in plasma was assayed by LC-MS/MS. The lower limit of quantification (LLOQ) for plasma was 1.45 pmol/L. No non-compartmental PK analysis was performed.
Time Frame: 5, 30 Minutes and 1, 2, 4, 8 and 12 Hours Post-dose
Population: Because of the dosing periods where formoterol was present at concentrations greater than 5% of the Cmax data for 4 subjects was excluded. A dosing error resulted in the exclusion of 1 subject and 1 subject had all data excluded from PK evaluation due to the plasma drug concentrations in conflict with the recorded randomization.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- F12D: Formoterol fumarate 12 μg via DPI/Placebo via pMDI
Arm/Group | MFF10 | F12M | F12D
Number analyzed (Participants) | 32 | 31 | 30
pmol/L
  Pre-Dose (N count MFF=15,F12M=17,F12D=16) | 0 (0) | 0 (0) | 0 (0)
  5-10 minutes (N=16, 17, 17) | 13.1 (12.2) | 16.3 (18.6) | 18.56 (9.19)
  30 minutes - 2 hours (N=16,17,17) | 27.5 (12.2) | 24.7 (18.7) | 23.1 (11.08)
  2 hours - 4 hours (N= 16, 17, 17) | 22.4 (15.1) | 17.7 (10.5) | 17.4 (6.44)
  4 hours - 8 hours (N= 16, 17, 17) | 12.3 (8.07) | 11.0 (5.3) | 11.3 (4.42)
  8 hours - 12 hours (N= 16, 16, 17) | 7.74 (5.68) | 6.66 (5.7) | 6.83 (4.76)

6. Secondary Outcome: Urinary Excretion of Formoterol Following a Single Dose of Formoterol Fumarate Alone and in Combination With Mometasone Furoate Via the pMDI and Formoterol Fumarate Via the Dry Powder Inhaler (DPI)
Description: Unchanged racemic formoterol in urine was assayed by LC-MS/MS. The lower limit of quantification (LLOQ) for urine was 0.0174 nmol/L expressed as free base. The amounts of unchanged formoterol excreted in urine from 0 to 3 hours (Ae0-3) and from 0 to 12 hours post-dose (Ae0-12) were calculated from the formoterol concentrations in urine and the urine volumes using non-compartmental methods.
Time Frame: 0 to 3 hrs and 0-12 hrs
Population: The pharmacokinetic population which was modified by the exclusion of dosing periods where formoterol was present at a concentration in excess of 5% of the Cmax.Five subjects were excluded due to various reasons.
Measure: Least Squares Mean (90% Confidence Interval); unit: nmol
Arm/Group | MFF10 | F12M | F12D
Number analyzed (Participants) | 32 | 31 | 30
nmol
  Ae (0-3) nmol (N=15,17,17) | 0.31 [0.20 to 0.49] | 0.52 [0.33 to 0.80] | 0.42 [0.27 to 0.65]
  Ae (0-12) nmol (N=16,17,17) | 1.14 [0.81 to 1.59] | 1.50 [1.08 to 2.08] | 1.33 [0.96 to 1.85]

ADVERSE EVENTS:
Arm/Group | F12M | F12D | MFF10 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.